CLINICAL TRIAL: NCT06543303
Title: A Phase 2, Double-Masked, Randomized, Vehicle-controlled Trial Evaluating the Efficacy and Safety of Cevimeline Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Evaluation of BTV100 in Subjects With Dry Eye Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioTheraVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTV100-CS201
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-masked, randomized, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked investigational product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BTV100 Low dose (Experimental): 1% Cevimeline Ophthalmic Solution
  Interventions: Drug: BTV100 Low dose
- BTV100 Mid dose (Experimental): 2% Cevimeline Ophthalmic Solution
  Interventions: Drug: BTV100 Mid dose
- BTV High dose (Experimental): 4% Cevimeline Ophthalmic Solution
  Interventions: Drug: BTV100 High dose
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTV100 Low dose — 1% Cevimeline Ophthalmic Solution
  Arms: BTV100 Low dose
Drug: BTV100 Mid dose — 2% Cevimeline Ophthalmic Solution
  Arms: BTV100 Mid dose
Drug: BTV100 High dose — 4% Cevimeline Ophthalmic Solution
  Arms: BTV High dose
Drug: Placebo — Placebo
  Arms: Vehicle

SUMMARY:
This study will be a randomized, vehicle-controlled, double-masked, multiple-dose, parallel-group study to evaluate the efficacy, safety and tolerability of repeat dosing of Cevimeline Ophthalmic Solution compared to the vehicle in subjects with Dry Eye Disease (DED).

DETAILED DESCRIPTION:
At the screening visit/Visit 1 (Day 1 minus 14 days), subjects who are eligible according to the inclusion and exclusion criteria will begin a 14-day run-in period during which they will self-administer 1 drop of single-masked vehicle to each eye twice daily (BID), morning and evening (at least 6-hour interval). At the time of the screening visit/Visit 1, subjects will be instructed to discontinue all over the counter (OTC) and prescription topical ophthalmic medications except for the vehicle or study drug throughout the study.

At Baseline/Visit 2 (Day 1), subjects who continue fulfilling inclusion/exclusion criteria will be randomized to study drug or vehicle.

Approximately120 subjects will be randomized. Subjects will be randomized to one of the following 4 treatment groups. Following randomization, subjects being masked to treatment assignments will be instructed to self-administer 1 drop of investigational product (IP) into each eye twice daily, morning and evening (at least 6-hour interval). Subjects will be instructed to return to the clinic to be evaluated at Day 15 (Visit 3), Day 29 (Visit 4), Day 57 (Visit 5), and Day 85 (Visit 6).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older (regardless of gender).
2. Provide written informed consent.
3. Willing and able to follow instructions and be available for required study visits during the study.
4. Best Corrected Visual Acuity (BCVA) of 20/100 or better in both eyes.
5. Ongoing moderate to severe Dry Eye Disease (DED) supported by a previous clinical diagnosis or a self-reported history of subjective complaints for at least 6 months prior to the screening visit, and meet all the following criteria in at least one eye (the same eye) at Visit 1 and Visit 2:

Exclusion Criteria:

1. Known hypersensitivity or contraindication to the study drug or its components.
2. Within 28 days prior to the screening visit (Visit 1), have taken or used: Topical ophthalmic, dermatologic or systemic calcineurin inhibitor (e.g. cyclosporine and tacrolimus), including Restasis® (cyclosporine) and Cequa® (cyclosporine)
3. Current use of contact lenses or anticipated use during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Schirmer test | Day 85
  Change from baseline in unanesthetized Schirmer test of study eye

SECONDARY OUTCOMES:
Schirmer test | Day 15, 29, 57 and 85.
  Proportion of subjects with an increase in unanesthetized Schirmer of 10 mm or more for study eye

CONTACTS AND LOCATIONS:
Overall Officials: Mulan Lee, PhD, Study Director — BioTheraVision, Inc.
Locations (6):
- Australia (2):
  - Cataract and Eye Surgery Centre, Victoria, Doncaster East, Victoria
  - Sydney Eye Hospital, Sydney
- Taiwan (4):
  - Chang Gung Memorial Hospital-Kaohsiung Branch, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-LinKou Branch, Taoyuan District